CLINICAL TRIAL: NCT03997578
Title: Non-incised Papillae Surgical Approach (NIPSA) and Connective Tissue Graft Plus Enamel Matrix Derivated and Xenograft for the Treatment of Periodontal Defects: a Controlled Clinical Trial
Brief Title: Non-incised Papillae Surgical Approach (NIPSA) and Connective Tissue Graft Plus Emdogain for Periodontal Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Antonio José Ortiz Ruiz, MD, Professor and researcher, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEI 1864/2018 - CBE 100/2018
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Periodontitis; Periodontal Bone Loss; Periodontal; Lesion
MeSH Terms: conditions — Periodontitis; Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NIPSA (Active Comparator): Patients will be treated with only NIPSA technique.
  Interventions: Procedure: NIPSA (Non-incised papilla surgical approach)
- NIPSA plus Connective tissue graft (Experimental): Patients will be treated with NIPSA technique associated to a connective tissue graft.
  Interventions: Procedure: NIPSA plus connective tissue graft

INTERVENTIONS:
Procedure: NIPSA (Non-incised papilla surgical approach) — To access the defect, a single horizontal or oblique apical incision will be made in the mucosa located on the bony cortex, far from the marginal tissues and apically to the edge of the bony crest delimiting the defect. The incision will be extended mesiodistally as necessary to allow access to the defect and correct debridement of the granulation tissue. The tissue coronal to the incision will be raised full thickness, trying to maintain the preoperative papillae architecture intact. The granulation tissue and epithelium of the pocket will be eliminated. The affected root will be scaled and planed, and calculus eliminated. Once the defect will be debrided, the regenerative biomaterials will be applied. Then the incision line will be sutured by a double suture line to facilitate closing without tension: The first with internal horizontal mattress sutures to approximate the connective tissue of both edges of the mucosal incision, and the second with single interrupted sutures.
  Arms: NIPSA
Procedure: NIPSA plus connective tissue graft — In these patients, the following methodology will be added to the technique described for the NIPSA group: once the biomaterials are applied, a connective tissue graft, taken at the level of the first upper molar, will be sutured to the base of the soft supra-alveolar tissue and to the palatal tissue, which has not been disinserted, using simple sutures.
  Arms: NIPSA plus Connective tissue graft

SUMMARY:
The present study pretends to show the results of combining a modification of the Non-incised papillae surgical approach (NIPSA) attempting to improve the outcome in the treatment of teeth with advanced periodontal support loss.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with periodontitis.
* plaque index and bleeding index of < 30%.
* periodontal lesions with pocket probing depth > 5 mm.
* intrabony defect > 3 mm.
* intrabony defect configuration including a 1 and/or 2-wall component, always involving the buccal wall.

Exclusion Criteria:

* patients with systemic diseases that contraindicated treatment.
* third molars.
* teeth with incorrect endodontic or restorative treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth (PD) | 12 months
  Probing pocket depth will be assessed with a periodontal probe, measured in mm from the gingival margin to the bottom of the pocket.
Clinical attachment level (CAL) | 12 months
  Clinical attachment level will be assessed with a periodontal probe, measured in mm from the cementoenamel junction (CEJ) to the bottom of the pocket.
Recession (REC) | 12 months
  Recession, will be assessed with a periodontal probe, measured in mmm on the buccal aspect, from the CEJ to the gingival margin zenith.
Location of the tip of the papillae (TP) | 12 months
  Location of the tip of the papillae. Taking as reference the level of the mid-axis of the tooth, will be measured the distance from the CEJ at the zenith of the tooth to the tip of the papilla. A positive value will be recorded when the tip of the papillae is located coronally to the CEJ and a negative value otherwise.
  This outcome will be assessed with a periodontal probe and measured in mmm.
Keratinized tissue width (KT) | 12 months
  Keratinized tissue width will be assessed with a periodontal probe, measured in mm on the buccal aspect, from the gingival margin to the mucogingival line.
Bleeding on probing | 12 months
  Bleeding on probing could be positive or negative.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Odontologico Del Sureste Slp, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreno Rodriguez JA, Ortiz Ruiz AJ, Caffesse RG. Supra-alveolar attachment gain in the treatment of combined intra-suprabony periodontal defects by non-incised papillae surgical approach. J Clin Periodontol. 2019 Sep;46(9):927-936. doi: 10.1111/jcpe.13158. Epub 2019 Jul 22. PMID 31190409
- [Background] Moreno Rodriguez JA, Ortiz Ruiz AJ, Caffesse RG. Periodontal reconstructive surgery of deep intraosseous defects using an apical approach. Non-incised papillae surgical approach (NIPSA): A retrospective cohort study. J Periodontol. 2019 May;90(5):454-464. doi: 10.1002/JPER.18-0405. Epub 2018 Nov 28. PMID 30421495